CLINICAL TRIAL: NCT01813409
Title: American College of Rheumatology Clinical Registry
Brief Title: Rheumatology Clinical Registry
Acronym: RCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American College of Rheumatology (Other)
Responsible Party: Sponsor
Other Study IDs: ACR-RCR
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The ACR Rheumatology Clinical Registry (RCR) is a tool developed to assist members in practice improvement, local population management, and efficient, successful participation in national quality programs. RCR integrates evidence-based quality measures aimed at improving care and drug safety for patients with rheumatoid arthritis, osteoarthritis, osteoporosis, gout and juvenile idiopathic arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Rheumatoid Arthritis

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Rheumatology patients
Sampling Method: Non-Probability Sample
Enrollment: 820 (Estimated)
Dates: Start 2009-08; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Quality of the treatment of rheumatoid arthritis and other diseases | Up to a year

SECONDARY OUTCOMES:
Submission to federal reporting programs | Up to a year

CONTACTS AND LOCATIONS:
Locations (1):
- Registry Site, Atlanta, Georgia, United States